CLINICAL TRIAL: NCT01717638
Title: A Phase 3, Open Label, Multi-Center, Extension Study to Assess Antibody Persistence and Response to a Third or Fifth Dose of Novartis Meningococcal B Recombinant Vaccine in 4-Year-Old Children Who Previously Participated in Study V72P12E1
Brief Title: Persistence of Antibody Levels and Response to Fifth or Third Meningococcal B Recombinant Vaccine in 4-year Old Healthy Children Who Previously Participated in Study V72P12E1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72P12E2; 2011-004931-30 (EudraCT Number)
Record Dates: First submitted 2012-10-18; First posted 2012-10-30 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningococcal disease, vaccines, children, persistence
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (13):
- B+R246_12_48 (Experimental): Previously received rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine + routine vaccines at 2, 4 and 6 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 12 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B+R246_18_48 (Experimental): Previously received rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine + routine vaccines at 2, 4 and 6 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 18 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B+R246_24_48 (Experimental): Previously received rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine + routine vaccines at 2, 4 and 6 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 24 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B246_12_48 (Experimental): Previously received 3 doses of rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine at 2, 4 and 6 months of age and routine vaccines at 3, 5 and 7 months of age, followed by a booster dose of rMenB+OMV NZ vaccine at 12 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B246_18_48 (Experimental): Previously received 3 doses of rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine at 2, 4 and 6 months of age and routine vaccines at 3,5 and 7 months of age, followed by a booster dose of rMenB+OMV NZ at 18 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B246_24_48 (Experimental): Previously received 3 doses of rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine at 2, 4 and 6 months of age and routine vaccines at 3, 5 and 7 months of age, followed by a booster dose of rMenB+OMV NZ vaccine at 24 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B+R234_12_48 (Experimental): Previously received 3 doses of rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine + routine vaccines at 2, 3 and 4 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 12 months of age. All subjects received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B+R234_18_48 (Experimental): Previously received rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine + routine vaccines at 2, 3 and 4 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 18 months of age. All subjects received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B+R234_24_48 (Experimental): Previously received rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine + routine vaccines at 2, 3 and 4 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 24 months of age. All subjects received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B12 14_48 (Experimental): Previously received two catch-up doses of rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine at 12 and14 months of age. All subjects received a 3rd dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B18 20_48 (Experimental): Previously received two catch-up doses of rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine at 18 & 20 months of age. All subjects received a 3rd dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B24 26_48 (Experimental): Previously received two catch-up doses of rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine at 24 & 26 months of age. All subjects received a 3rd dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
  Interventions: Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine
- B48_50 (Experimental): Newly recruited 4 year old naive subjects who received 2 catch-up doses of rMenB+OMV NZ, ie, Meningococcal (group B) multicomponent recombinant adsorbed vaccine, two months apart, in the present study.
  Interventions: Biological: 2 doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine

INTERVENTIONS:
Biological: 1 dose of Meningococcal (group B) multicomponent recombinant adsorbed vaccine — 0.5 mL of Meningococcal (group B) multicomponent recombinant adsorbed vaccine, Intramuscular, single dose
  Other Names: rMenB+OMV NZ
  Arms: B+R234_12_48; B+R234_18_48; B+R234_24_48; B+R246_12_48; B+R246_18_48; B+R246_24_48; B12 14_48; B18 20_48; B24 26_48; B246_12_48; B246_18_48; B246_24_48
Biological: 2 doses of Meningococcal (group B) multicomponent recombinant adsorbed vaccine — 0.5 mL of Meningococcal (group B) multicomponent recombinant adsorbed vaccine, Intramuscular, two doses, two months apart
  Other Names: rMenB+OMV NZ
  Arms: B48_50

SUMMARY:
It is a Phase 3 extension of study V72P12E1 (NCT00944034). The main aim of the second extension study is to explore the bactericidal antibody persistence in 4-year-old children after a fourth dose boost of rMenB+OMV NZ or after a two-dose catch-up schedule of rMenB+OMV NZ administered to toddlers as part of their respective vaccination courses in study V72P12E1.

In addition, this study will characterize the antibody response to a fifth dose boost in all children who received a three-dose primary series of rMenB+OMV NZ at 2, 3, 4 months of age (in parent study V72P12, NCT00721396), and only in a subset of children who received a three-dose primary series of rMenB+OMV NZ at 2, 4, 6 months of age (in parent study V72P12). Antibody response will also be characterized to a third dose boost of rMenB+OMV NZ administered at approximately 4 years of age in all children who received a two catch-up doses of rMenB+OMV NZ as toddlers in study V72P12E1.

Finally, the safety and immunogenicity of two catch-up doses of rMenB+OMV NZ administered 2 months apart to healthy naïve children at 4 years of age will be assessed.

ELIGIBILITY:
Inclusion Criteria:

A. Inclusion Criteria for naïve subjects, newly enrolled (B48_50):

1. 4 years old (48 to 60 months) healthy male and female subjects will be recruited from the same sites as in study V72P12E1. The age window is defined as the first day the subject turns 4 years old up to the day before the subject turns 5 years old.
2. For whom parent/legal guardian(s) has given written informed consent after the nature of the study has been explained.
3. For whom parent/legal guardian(s) confirmed availability for the visit(s) scheduled in the study.
4. In good health as determined by medical history, physical examination, clinical judgment of the investigator.

B. Inclusion Criteria for follow-on participants (Groups B+R246 12_48, B+R246 18_48, B+R246 24_48, B246 12_48, B246 18_48, B246 24_48, B+R234 12_48, B+R234 18_48, B+R234 24_48, B12 14_48, B18 20_48, B24 26_48):

Inclusion criteria are the same as for Group B48_50, with the addition that they are subjects who completed the vaccination course of V72P12E1 study.

Exclusion Criteria:

A. Exclusion Criteria for naïve subjects, newly enrolled (Group 7):

1. Subjects whose parents/legal guardians are unwilling or unable to give written informed consent to participate in the study.
2. History of any meningococcal B vaccine administration.
3. Previous ascertained or suspected disease caused by N. meningitidis.
4. Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis.
5. History of allergic reaction to any vaccine component.
6. Significant chronic infection.
7. Any serious chronic or progressive disease according to the judgment of the investigator (e.g., neoplasm, diabetes mellitus Type I, cardiac disease, hepatic disease, progressive neurological disease or seizure, either associated with fever or as part of an underlying neurological disorder or syndrome, autoimmune disease, HIV infection or AIDS, or blood dyscrasias or diathesis, signs of cardiac or renal failure or severe malnutrition).
8. Known or suspected impairment/alteration of the immune system resulting from (for example) receipt of chronic immunosuppressive therapy or immunostimulants.
9. Participation in another clinical trial within 90 days prior to enrolment or planned for during study.
10. Family members and household members of research staff.
11. Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

B. Exclusion Criteria for follow-on participants ((Groups B+R246 12_48, B+R246 18_48, B+R246 24_48, B246 12_48, B246 18_48, B246 24_48, B+R234 12_48, B+R234 18_48, B+R234 24_48, B12 14_48, B18 20_48, B24 26_48):

Exclusion criteria are the same as for Group B48_50, with the exception of criterion 2 and excluding participation in V72P12E1 for criterion 9.

Ages: 48 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 805 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (29):
- Czechia (17):
  - Ordinace praktickeho lekare pro deti a dorost, Jaroměř, Alšova 466
  - Ordinace praktickeho lekare pro deti a dorost, Jaroměř, Dr. E.Beneše 191
  - Ordinace praktickeho lekare pro deti a dorost, Sezemice, Havlickova 168
  - Ordinace praktickeho lekare pro deti a dorost, Hronov, Hostovského 485
  - Ordinace praktickeho lekare pro deti a dorost, Česká Skalice, Husovo Namesti 36
  - Ordinace praktickeho lekare pro deti a dorost, Pardubice, L.Male 656
  - Ordinace praktickeho lekare pro deti a dorost, Hradec Králové, Manesova 646
  - Ordinace praktickeho lekare pro deti a dorost, Hronov, Palackeho 517
  - Ordinace praktickeho lekare pro deti a dorost, Hradec Králové, Pardubicka 752
  - Ordinace praktickeho lekare pro deti a dorost, Chlumec nad Cidlinou, Pernstynska 127/i
  - Nemocnice Náchod, Náchod, Purkynova 446
  - Ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec, Ruských Legií 352
  - Ordinace praktickeho lekare pro deti a dorost, Pardubice, Sladkovskeho 2617
  - Ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec, Sídliste Vajgar 724/iii
  - Fakulta vojenskeho zdravotnictvi UO, Hradec Králové, Trebesska 1575
  - Ordinace praktickeho lekare pro deti a dorost, Holice, U Kaplicky 1042
  - Ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec, U nemocnice380/III
- Italy (4):
  - Universita di Firenze -Pediatria, Florence
  - IRCCS Cà Granda, Milan
  - Ospedale Maggiore della Carita, Novara
  - Dip Pediatria AO Padova, Padua
- Spain (4):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela A Coruña
  - Hospital Universitario Dr. Peset, Valencia
  - Centro Superior de Investigacion en Salud Publica/Clinica Universitaria San Vicente Martir, Valencia
  - Complexo Hospitalario Xeral Cies, Vigo Pontevedra
- United Kingdom (4):
  - Oxford Vaccine Group - Centre for Clinical Vaccinology and Tropical Medicine Churchill Hospital, Oxford, Headington
  - North Bristol NHS Trust, Bristol
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - St Georges Hospital, London

REFERENCES:
- [Derived] Sadarangani M, Sell T, Iro MA, Snape MD, Voysey M, Finn A, Heath PT, Bona G, Esposito S, Diez-Domingo J, Prymula R, Odueyungbo A, Toneatto D, Pollard AJ; European MenB Vaccine Study Group. Persistence of immunity after vaccination with a capsular group B meningococcal vaccine in 3 different toddler schedules. CMAJ. 2017 Oct 16;189(41):E1276-E1285. doi: 10.1503/cmaj.161288. PMID 29038320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 4 centers from the UK, 4 centers from Italy, 4 centers from Spain, 19 centers from Czech Republic.
Pre-assignment Details: All subjects were included in the trial.
Groups:
- B+R246_12_48: Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 4 and 6 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 12 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B+R246_18_48: Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 4 and 6 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 18 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B+R246_24_48: Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 4 and 6 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 24 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B246_12_48: Previously received 3 doses of rMenB+OMV NZ vaccine at 2, 4 and 6 months of age and routine vaccines at 3, 5 and 7 months of age, followed by a booster dose of rMenB+OMV NZ vaccine at 12 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B246_18_48: Previously received 3 doses of rMenB+OMV NZ vaccine at 2, 4 and 6 months of age and routine vaccines at 3,5 and 7 months of age, followed by a booster dose of rMenB+OMV NZ at 18 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B246_24_48: Previously received 3 doses of rMenB+OMV NZ vaccine at 2, 4 and 6 months of age and routine vaccines at 3, 5 and 7 months of age, followed by a booster dose of rMenB+OMV NZ at 24 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B+R234_12_48: Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 3 and 4 months of age followed by a booster dose of rMenB+OMV NZ at 12months of age. All subjects received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B+R234_18_48: Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 3 and 4 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 18months of age. All subjects received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B+R234_24_48: Previously received rMenB+OMV NZ vaccine + routine vaccines at 2, 3 and 4 months of age followed by a booster dose of rMenB+OMV NZ vaccine at 24 months of age. All subjects received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B12 14_48: Previously received two catch-up doses of rMenB+OMV NZ vaccine at 12 &14 months of age. All subjects received a 3rd dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B18 20_48: Previously received two catch-up doses of rMenB+OMV NZ vaccine at 18 & 20 months of age. All subjects received a 3rd dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B24 26_48: Previously received two catch-up doses of rMenB+OMV NZ vaccine at 24 & 26 months of age. All subjects received a 3rd dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B48_50: Newly recruited 4 year old naive subjects who received 2 catch-up doses of rMenB+OMV NZ vaccine, two months apart, in the present study.
Period: Overall Study
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48 | B12 14_48 | B18 20_48 | B24 26_48 | B48_50
Started | 67 | 61 | 60 | 66 | 64 | 55 | 43 | 29 | 28 | 100 | 11 | 12 | 209
Completed | 67 | 60 | 59 | 66 | 63 | 54 | 41 | 28 | 26 | 99 | 11 | 12 | 190
Not Completed | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 19
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Father in hospital | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 18

BASELINE CHARACTERISTICS:
Population: Anaysis was done on the all enrolled population, ie, all subjects who have signed an informed consent, undergone screening procedure(s) and were randomized.
Groups:
- B48 50: Newly recruited 4 year old naive subjects who received 2 catch-up doses of rMenB+OMV NZ vaccine, two months apart, in the present study.
- Total: Total of all reporting groups
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48 | B12 14_48 | B18 20_48 | B24 26_48 | B48 50 | Total
Number analyzed (Participants) | 67 | 61 | 60 | 66 | 64 | 55 | 43 | 29 | 28 | 100 | 11 | 12 | 209 | 805
Age, Continuous [Mean (Standard Deviation); unit: Months] | 51.8 (3.4) | 52.1 (3.4) | 51.7 (3.5) | 51.7 (3.5) | 51.3 (3.7) | 52.3 (3.7) | 51.8 (3.4) | 51.4 (3.4) | 53.1 (3.5) | 51.7 (3.3) | 53.4 (4.3) | 56.8 (1.5) | 53.7 (3.6) | 52.4 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 33 | 28 | 32 | 30 | 24 | 17 | 13 | 50 | 6 | 4 | 99 | 387
  Male | 44 | 33 | 27 | 38 | 32 | 25 | 19 | 12 | 15 | 50 | 5 | 8 | 110 | 418

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Persisting Serum Bactericidal Titers ≥1:5 and ≥1:8 (at 4 Years of Age), Who Had Previously Received Three Primary Doses and One Booster Dose of rMenB+OMV NZ Vaccine According to Different Schedules
Description: The antibody persistence at 4 years of age in children who had previously received 3 primary doses (at 2, 3, 4, or 2, 4, 6 months) followed by a booster dose (at 12,18 or 24 months) of rMenB+OMV NZ vaccine according to different schedules is compared with the response in naïve children and reported as percentages of subjects with human serum bactericidal assay (hSBA) titers ≥1:5 and ≥1:8.
  The functional bactericidal antibodies directed against serogroup B meningococci were assessed using the Serum Bactericidal Assay (SBA) using human serum as the source of exogenous complement (hSBA).
Time Frame: Day 1 (24-36 months post booster; baseline for naive)
Population: Full Analysis Set (Fas), Persistency: All subjects in the enrolled population who provided at least one evaluable serum sample at baseline (visit 1). Persistence data sets include nonvaccination and vaccination subsets of subjects from different groups with different primary vaccination schedules of MenB+Routine vaccines and routine vaccines.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- B246_12_48: Previously received 3 doses of rMenB+OMV NZ vaccine at 2, 4 and 6 months of age and routine vaccines at 3,5 and 7 months of age, followed by a booster dose of rMenB+OMV NZ vaccine at 12 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B246_24_48: Previously received 3 doses of rMenB+OMV NZ vaccine at 2, 4 and 6 months of age and routine vaccines at 3,5 and 7 months of age, followed by a booster dose of rMenB+OMV NZ at 24 months of age. One third of subjects from this group received a 5th dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48 | B48 50
Number analyzed (Participants) | 67 | 60 | 60 | 66 | 63 | 54 | 42 | 28 | 28 | 206
Percentages of subjects
  H44/76 - ≥1:5; N=67,60,59,65,63,54,42,28,28,206 | 12 [5 to 22] | 18 [10 to 30] | 24 [14 to 37] | 20 [11 to 32] | 27 [17 to 40] | 35 [23 to 49] | 12 [4 to 26] | 25 [11 to 45] | 21 [8 to 41] | 0 [0 to 3]
  5/99 - ≥1:5; N=67,60,58,64,62,54,42,28,28,200 | 93 [83 to 98] | 98 [91 to 100] | 97 [88 to 100] | 97 [89 to 100] | 100 [94 to 100] | 100 [93 to 100] | 90 [77 to 97] | 89 [72 to 98] | 96 [82 to 100] | 5 [2 to 8]
  NZ 98/254 - ≥ 1:5 | 9 [3 to 18] | 8 [3 to 18] | 12 [5 to 23] | 9 [3 to 19] | 11 [5 to 22] | 9 [3 to 20] | 10 [3 to 23] | 11 [2 to 28] | 11 [2 to 28] | 0 [0 to 3]
  M10713 - ≥1:5; N=65,59,58,62,60,54,40,28,28,192 | 54 [41 to 66] | 68 [54 to 79] | 74 [61 to 85] | 55 [42 to 68] | 53 [40 to 66] | 80 [66 to 89] | 68 [51 to 81] | 75 [55 to 89] | 75 [55 to 89] | 60 [53 to 67]
  H44/76-≥1:8; N=67,60,59,65,63,54,42,28,28,206 | 7 [2 to 17] | 10 [4 to 21] | 17 [8 to 29] | 11 [4 to 21] | 24 [14 to 36] | 28 [16 to 42] | 7 [1 to 19] | 21 [8 to 41] | 21 [8 to 41] | 0 [0 to 3]
  5/99 - ≥1:8; N=67,60,58,64,62,54,42,28,28,200 | 91 [82 to 97] | 97 [88 to 100] | 93 [83 to 98] | 94 [85 to 98] | 94 [84 to 98] | 100 [93 to 100] | 90 [77 to 97] | 86 [67 to 96] | 96 [82 to 100] | 3 [1 to 6]
  NZ 98/254 - ≥ 1:8 | 4 [1 to 13] | 5 [1 to 14] | 8 [3 to 18] | 8 [3 to 17] | 3 [0 to 11] | 4 [0 to 13] | 2 [0.06 to 13] | 7 [1 to 24] | 11 [2 to 28] | 0 [0 to 3]
  M10713 - ≥1:8; N=65,59,58,62,60,54,40,28,28,192 | 49 [37 to 62] | 53 [39 to 66] | 60 [47 to 73] | 48 [35 to 61] | 45 [32 to 58] | 65 [51 to 77] | 60 [43 to 75] | 61 [41 to 78] | 61 [41 to 78] | 56 [48 to 63]

2. Primary Outcome: Persisting Antibody Titers in Children (at 4 Years of Age) Who Had Previously Received Three Primary Doses and One Booster Dose of rMenB+OMV NZ Vaccine According to Different Schedules
Description: The persisting antibody titers at 4 years of age in children who had previously received 3 primary doses (at 2, 3, 4, or 2, 4, 6 months) followed by a booster dose (at 12, 18 or 24 months) of rMenB+OMV NZ vaccine according to different schedules is compared with the titers in naive children and reported as geometric mean titers (GMTs).
Time Frame: Day 1 (24-36 months post booster; baseline for naive)
Population: FAS, Persistency.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48 | B48 50
Number analyzed (Participants) | 67 | 60 | 60 | 66 | 63 | 54 | 42 | 28 | 28 | 206
Titers
  H44/76; N=67,60,59,65,63,54,42,28,28,206 | 1.75 [1.36 to 2.25] | 1.68 [1.29 to 2.19] | 2.41 [1.83 to 3.19] | 1.72 [1.29 to 2.29] | 1.99 [1.49 to 2.65] | 2.69 [1.96 to 3.7] | 1.51 [1.04 to 2.18] | 2.2 [1.38 to 3.49] | 2.2 [1.37 to 3.53] | 1.04 [1.01 to 1.07]
  5/99; N=67,60,58,64,62,54,42,28,28,200 | 36 [27 to 48] | 69 [50 to 94] | 69 [50 to 96] | 59 [45 to 78] | 57 [43 to 75] | 111 [82 to 151] | 52 [34 to 81] | 62 [36 to 108] | 101 [57 to 177] | 1.15 [1.05 to 1.27]
  NZ 98/254 | 1.25 [1.03 to 1.52] | 1.29 [1.05 to 1.59] | 1.38 [1.11 to 1.72] | 1.48 [1.2 to 1.83] | 1.34 [1.08 to 1.66] | 1.52 [1.2 to 1.92] | 1.32 [1.05 to 1.65] | 1.25 [0.94 to 1.66] | 1.62 [1.21 to 2.16] | 1.01 [0.99 to 1.03]
  M10713; N=65,59,58,62,60,54,40,28,28,192 | 6.14 [4.19 to 8.99] | 7.36 [4.94 to 11] | 9.08 [5.97 to 14] | 7.86 [5.17 to 12] | 7.77 [5.07 to 12] | 15 [9.49 to 24] | 9.61 [5.81 to 16] | 11 [5.92 to 20] | 11 [5.9 to 21] | 8.75 [6.74 to 11]

3. Primary Outcome: Geometric Mean Ratios (GMRs) in Children (at 4 Years of Age) Who Had Previously Received Three Primary Doses and One Booster Dose of rMenB+OMV NZ Vaccine According to Different Schedules
Description: The GMRs of GMTs (48 months/one month post booster vaccination) at 4 years of age in children who had previously received 3 primary doses (at 2, 3, 4, or 2, 4, 6 months) followed by a booster dose (at 12,18 or 24 months) of rMenB+OMV NZ vaccine according to different schedules is reported.
Time Frame: Day 1 (24-36 months post booster dose; baseline for naive)
Population: FAS, Persistency.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48
Number analyzed (Participants) | 63 | 57 | 54 | 59 | 56 | 47 | 39 | 28 | 25
Ratio
  H44/76; N=62,56,52,57,55,46,38,27,25,206 | 0.012 [0.0091 to 0.017] | 0.013 [0.0096 to 0.018] | 0.023 [0.016 to 0.033] | 0.0092 [0.0066 to 0.013] | 0.013 [0.0097 to 0.018] | 0.023 [0.016 to 0.033] | 0.0091 [0.0064 to 0.013] | 0.023 [0.015 to 0.036] | 0.023 [0.014 to 0.036]
  5/99; N=61,57,50,57,55,44,37,27,25,200 | 0.029 [0.023 to 0.037] | 0.032 [0.026 to 0.041] | 0.043 [0.033 to 0.056] | 0.031 [0.024 to 0.041] | 0.034 [0.026 to 0.045] | 0.054 [0.04 to 0.074] | 0.035 [0.026 to 0.048] | 0.037 [0.025 to 0.054] | 0.055 [0.037 to 0.081]
  NZ 98/254 | 0.028 [0.021 to 0.039] | 0.094 [0.067 to 0.13] | 0.071 [0.05 to 0.1] | 0.043 [0.031 to 0.06] | 0.081 [0.058 to 0.11] | 0.11 [0.075 to 0.16] | 0.03 [0.02 to 0.044] | 0.082 [0.05 to 0.14] | 0.066 [0.038 to 0.11]
  M10713; N=26,24,25 | NA [NA to NA] — GMTs were not calculated for this group in the parent study therefore the ratios cannot be available. | NA [NA to NA] — GMTs were not calculated for this group in the parent study therefore the ratios cannot be available. | NA [NA to NA] — GMTs were not calculated for this group in the parent study therefore the ratios cannot be available. | NA [NA to NA] — GMTs were not calculated for this group in the parent study therefore the ratios cannot be available. | NA [NA to NA] — GMTs were not calculated for this group in the parent study therefore the ratios cannot be available. | NA [NA to NA] — GMTs were not calculated for this group in the parent study therefore the ratios cannot be available. | 0.67 [0.32 to 1.4] | 0.91 [0.4 to 2.05] | 0.47 [0.21 to 1.07]

4. Secondary Outcome: Percentages of Subjects With Persisting Serum Bactericidal Titers ≥1:5 and ≥1:8 (at 4 Years of Age), Who Had Previously Received Two Catch up Doses of rMenB+OMV NZ Vaccine According to Different Schedules
Description: The antibody persistence in children at 4 year of age, who had previously received 2 catch up doses (at 12, 14 or 18, 20 or 24, 26 months) according to different schedules is reported as percentages of subjects with hSBA titers ≥1:5 and hSBA titers ≥1:8.
Time Frame: Day 1 (22-34 months post last MenB vaccine)
Population: FAS, Persistency. Note: Reporting groups in this endpoint and in endpoints 5 and 6 received vaccination according to different schedules with respect to the groups reported in endpoints 1, 2 and 3.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- B12 14_48: Previously received routine vaccines at 2,4 and 6 months of age, followed by two catch-up doses of rMenB+OMV NZ vaccine at 12 &14 months of age. All subjects received a 3rd dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B18 20_48: Previously received two catch-up doses of rMenB+OMV NZ vaccine at 18 & 20 months of age. All subjects from this group received a 3rd dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
- B24 26_48: Previously received two catch-up doses of rMenB+OMV NZ vaccine at 24 & 26 months of age. All subjects from this group received a 3rd dose of rMenB+OMV NZ vaccine in the present study at 4 years of age.
Arm/Group | B12 14_48 | B18 20_48 | B24 26_48 | B48 50
Number analyzed (Participants) | 96 | 11 | 11 | 206
Percentages of subjects
  hSBA≥ 1:5 (H44/76 strain) | 11 [6 to 20] | 9 [0 to 41] | 9 [0 to 41] | 0 [0 to 3]
  hSBA≥ 1:5 (5/99 strain; N=96,11,11,200) | 84 [76 to 91] | 100 [72 to 100] | 100 [72 to 100] | 5 [2 to 8]
  hSBA≥ 1:5 (NZ 98/254 strain) | 3 [1 to 9] | 18 [2 to 52] | 0 [0 to 28] | 0 [0 to 3]
  hSBA≥ 1:5 (M10713 strain; N=96,10,10,192) | 59 [49 to 69] | 60 [26 to 88] | 60 [26 to 88] | 60 [53 to 67]
  hSBA≥ 1:8 (H44/76 strain) | 8 [4 to 16] | 9 [0 to 41] | 0 [0 to 28] | 0 [0 to 3]
  hSBA≥ 1:8 (5/99 strain; N=96,11,11,200) | 81 [72 to 88] | 100 [72 to 100] | 100 [72 to 100] | 3 [1 to 6]
  hSBA≥ 1:8 (NZ 98/254 strain) | 2 [0 to 7] | 18 [2 to 52] | 0 [0 to 28] | 0 [0 to 3]
  hSBA≥ 1:8 (M10713 strain; N=96,10,10,192) | 49 [39 to 59] | 40 [12 to 74] | 60 [26 to 88] | 56 [48 to 63]

5. Secondary Outcome: Persisting Antibody Titers in Children (at 4 Years of Age) Who Had Previously Received Two Catch up Doses of rMenB+OMV NZ Vaccine According to Different Schedules
Description: The persisting GMTs in children at 4 years of age, who had previously received 2 catch up doses (at 12, 14 or 18, 20 or 24, 26 months) of rMenB+OMV NZ vaccine according to different schedules are reported.
Time Frame: Day 1 (22-36 months post last MenB vaccine; baseline for naive)
Population: FAS, Persistency.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B12 14_48 | B18 20_48 | B24 26_48 | B48 50
Number analyzed (Participants) | 96 | 11 | 11 | 206
Titers
  H44/76 strain | 1.61 [1.3 to 2] | 2.03 [1.11 to 3.72] | 1.69 [0.91 to 3.12] | 1.04 [1.01 to 1.07]
  5/99 strain; N=96, 11, 11, 200 | 23 [17 to 32] | 47 [20 to 112] | 69 [29 to 165] | 1.15 [1.05 to 1.27]
  NZ 98/254 strain | 1.15 [0.96 to 1.37] | 2.68 [1.65 to 4.36] | 1.06 [0.65 to 1.75] | 1.01 [0.99 to 1.03]
  M10713 strain; N=96, 10, 10, 192 | 7.83 [5.54 to 11] | 9.67 [3.54 to 26] | 8.4 [3.03 to 23] | 8.75 [6.74 to 11]

6. Secondary Outcome: GMRs of GMTs in Children (at 4 Years of Age) Who Had Previously Received Two Catch up Doses of rMenB+OMV NZ Vaccine According to Different Schedules
Description: The GMRs of GMTs (48 months/one month post last vaccination) in children at 4 years of age who had previously received 2 catch up doses (at 12, 14 or 18, 20 or 24, 26 months) of rMenB+OMV NZ vaccine according to different schedules.
Time Frame: Day 1 (22-34 months post last MenB vaccine)
Population: FAS, Persistency.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | B12 14_48 | B18 20_48 | B24 26_48
Number analyzed (Participants) | 88 | 9 | 10
Ratio
  H44/76 strain | 0.092 [0.069 to 0.12] | 0.18 [0.078 to 0.43] | 0.2 [0.086 to 0.45]
  5/99 strain | 0.45 [0.34 to 0.59] | 1.9 [0.84 to 4.29] | 1.36 [0.62 to 3]
  NZ 98/254 strain; N=88, 9, 8 | 0.28 [0.21 to 0.37] | 0.73 [0.32 to 1.68] | 0.42 [0.17 to 1.01]
  M10713 strain; N=7, 7, 8 | 11 [3.34 to 38] | 6.05 [1.45 to 25] | 6.88 [1.68 to 28]

7. Secondary Outcome: Percentages of Subjects With Serum Bactericidal Titers ≥1:5 and ≥1:8 After a 5th Dose of rMenB+OMV NZ Vaccine (at 4 Years of Age) Who Had Previously Received 3 Primary Doses and a Booster Dose of the Same Vaccine According to Different Schedules
Description: The Percentages of subjects with hSBA titers ≥1:5 and ≥1:8, one month after a 5th dose of rMenB+OMV NZ vaccine was given children who had previously received 3 primary doses (at 2, 3, 4,or 2, 4, 6 months) and a booster dose (at 12, 18 or 24 months) of the same vaccine according to different schedules is compared with the hSBA response of children who received first dose of rMenB+OMV NZ at 4 years of age.
Time Frame: Day 31 (1 month post vaccination)
Population: Analysis was done on FAS, Immunogenicity, ie, all subjects in the enrolled population who actually received a study vaccination, and provided at least one evaluable serum sample at post baseline.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48 | B48 50
Number analyzed (Participants) | 26 | 18 | 16 | 16 | 26 | 15 | 40 | 26 | 26 | 175
Percentages of subjects
  H44/76 - ≥1:5; N=26,18,16,16,26,15,39,26,26,175 | 100 [87 to 100] | 100 [81 to 100] | 100 [79 to 100] | 100 [79 to 100] | 100 [87 to 100] | 100 [78 to 100] | 97 [87 to 100] | 100 [87 to 100] | 100 [87 to 100] | 71 [64 to 78]
  5/99 - ≥1:5; N=26,18,16,16,26,15,38,26,26,171 | 100 [87 to 100] | 100 [81 to 100] | 100 [79 to 100] | 100 [79 to 100] | 100 [87 to 100] | 100 [78 to 100] | 100 [91 to 100] | 100 [87 to 100] | 100 [87 to 100] | 90 [85 to 94]
  NZ 98/254 - ≥1:5; N=26,18,16,16,26,15,40,26,26,173 | 92 [75 to 99] | 83 [59 to 96] | 94 [70 to 100] | 81 [54 to 96] | 88 [70 to 98] | 80 [52 to 96] | 95 [83 to 99] | 92 [75 to 99] | 92 [75 to 99] | 24 [18 to 31]
  M10713 - ≥1:5; N=25,18,16,14,25,15,36,25,25,167 | 84 [64 to 95] | 89 [65 to 99] | 88 [62 to 98] | 93 [66 to 100] | 96 [80 to 100] | 93 [68 to 100] | 97 [85 to 100] | 100 [86 to 100] | 100 [86 to 100] | 77 [70 to 83]
  H44/76 - ≥1:8; N=26,18,16,16,26,15,39,26,26,175 | 96 [80 to 100] | 100 [81 to 100] | 100 [79 to 100] | 100 [79 to 100] | 96 [80 to 100] | 100 [78 to 100] | 97 [87 to 100] | 100 [87 to 100] | 96 [80 to 100] | 63 [55 to 70]
  5/99 - ≥1:8; N=26,18,16,16,26,15,38,26,26,171 | 100 [87 to 100] | 100 [81 to 100] | 100 [79 to 100] | 100 [79 to 100] | 100 [87 to 100] | 100 [78 to 100] | 100 [91 to 100] | 100 [87 to 100] | 100 [87 to 100] | 87 [81 to 92]
  NZ 98/254 - ≥1:8; N=26,18,16,16,26,15,40,26,26,173 | 85 [65 to 96] | 61 [36 to 83] | 81 [54 to 96] | 75 [48 to 93] | 88 [70 to 98] | 80 [52 to 96] | 88 [73 to 96] | 81 [61 to 93] | 88 [70 to 98] | 17 [12 to 24]
  M10713 - ≥1:8; N=25,18,16,14,25,15,36,25,25,167 | 76 [55 to 91] | 89 [65 to 99] | 88 [62 to 98] | 93 [66 to 100] | 96 [80 to 100] | 93 [68 to 100] | 97 [85 to 100] | 100 [86 to 100] | 96 [80 to 100] | 74 [67 to 81]

8. Secondary Outcome: GMTs in Children Following a Fifth Dose of rMenB+OMV NZ Vaccine (at 4 Years of Age) Who Had Previously Received 3 Primary Doses and a Booster Dose of the Same Vaccine According to Different Schedules
Description: The GMTs, at one month after a 5th dose of rMenB+OMV NZ vaccine in children who had previously received 3 primary doses (at 2, 3, 4, or 2, 4, 6 months) and a booster dose (at 12, 18 or 24 months) of rMenB+OMV NZ vaccine according to different schedules, are compared with the GMTs of children who received first dose of rMenB+OMV NZ at 4 years of age.
Time Frame: Day 31 (1 month post vaccination)
Population: Analysis was done on FAS (Immunogenicity).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48 | B48 50
Number analyzed (Participants) | 26 | 18 | 16 | 16 | 26 | 15 | 40 | 26 | 26 | 175
Titers
  H44/76 strain; N=26,18,16,16,26,15,39,26,26,175 | 108 [70 to 168] | 115 [68 to 195] | 107 [61 to 188] | 173 [98 to 303] | 191 [123 to 297] | 212 [119 to 379] | 167 [109 to 258] | 146 [85 to 251] | 135 [78 to 235] | 11 [8.51 to 14]
  5/99 strain; N=26,18,16,16,26,15,38,26,26,171 | 754 [478 to 1190] | 1719 [993 to 2976] | 933 [518 to 1682] | 1959 [1091 to 3517] | 1387 [878 to 2191] | 1954 [1068 to 3575] | 1711 [1186 to 2470] | 1239 [787 to 1953] | 1280 [803 to 2041] | 34 [27 to 42]
  NZ 98/254 strain; N=26,18,16,16,26,15,40,26,26,173 | 22 [13 to 36] | 11 [5.66 to 20] | 28 [14 to 55] | 16 [8.2 to 31] | 21 [13 to 36] | 15 [7.66 to 31] | 26 [18 to 36] | 18 [12 to 28] | 27 [18 to 42] | 2.25 [1.84 to 2.75]
  M10713 strain; N=25,18,16,14,25,15,36,25,25,167 | 22 [13 to 37] | 19 [10 to 36] | 28 [14 to 54] | 32 [16 to 65] | 37 [22 to 63] | 33 [17 to 64] | 53 [40 to 71] | 58 [40 to 84] | 51 [35 to 73] | 20 [15 to 25]

9. Secondary Outcome: Geometric Mean Ratios of GMTs in Subjects Following a Fifth Dose of rMenB+OMV NZ Vaccine (at 4 Years of Age), Who Had Previously Received 3 Primary Doses and a Booster Dose of the Same Vaccine According to Different Schedules
Description: The GMRs of GMTs (one month post booster/48 months persistence), one month after a 5th dose of rMenB+OMV NZ vaccine was given children, who had previously received 3 primary doses (at 2, 3, 4, or 2, 4, 6 months) and a booster dose (at 12, 18 or 24 months) of rMenB+OMV NZ vaccine according to different schedules is compared with the GMR (one month post 1 dose\baseline) of children who received first dose of rMenB+OMV NZ at 4 years of age.
Time Frame: Day 31 (1 month post vaccination)
Population: Analysis was done on FAS (Immunogenicity).
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48 | B48 50
Number analyzed (Participants) | 26 | 18 | 16 | 16 | 26 | 15 | 40 | 25 | 26 | 175
Ratio
  H44/76 strain; N=26,18,16,16,26,15,39,25,26,175 | 60 [40 to 92] | 72 [44 to 120] | 41 [24 to 71] | 77 [45 to 132] | 88 [58 to 134] | 46 [26 to 80] | 109 [71 to 167] | 63 [37 to 108] | 64 [37 to 110] | 10 [8.2 to 13]
  5/99 strain; N=26,18,16,15,25,15,38,25,26,168 | 32 [22 to 47] | 23 [15 to 36] | 15 [9.45 to 25] | 30 [18 to 49] | 20 [13 to 29] | 18 [11 to 29] | 33 [23 to 49] | 20 [12 to 32] | 12 [7.16 to 19] | 29 [23 to 37]
  NZ 98/254 strain; N=26,18,16,16,26,15,40,25,26,173 | 17 [10 to 29] | 10 [5.43 to 19] | 19 [9.54 to 37] | 8.93 [4.57 to 17] | 17 [10 to 29] | 13 [6.48 to 26] | 19 [14 to 27] | 14 [9.35 to 22] | 17 [11 to 26] | 2.25 [1.84 to 2.75]
  M10713 strain; N=24,17,16,12,23,15,35,24,25,158 | 3.15 [1.81 to 5.48] | 4.46 [2.31 to 8.6] | 3.36 [1.69 to 6.7] | 3.49 [1.58 to 7.7] | 3.74 [2.12 to 6.59] | 4.21 [2.08 to 8.51] | 5.35 [3.48 to 8.21] | 3.86 [2.23 to 6.66] | 4.04 [2.35 to 6.94] | 2 [1.62 to 2.46]

10. Secondary Outcome: Percentages of Subjects With Fourfold Increase in hSBA Titers After Receiving a Fifth Dose of rMenB+OMV NZ Vaccine (at 4 Years of Age), Who Had Previously Received 3 Primary Doses and a Booster Dose of the Same Vaccine According to Different Schedules
Description: The fourfold increase in hSBA titers, one month after a 5th dose of rMenB+OMV NZ vaccine was given to children, who had previously received 3 primary doses (at 2, 3, 4, or 2, 4, 6 months) and a booster dose (at 12,18 or 24 months) of rMenB+OMV NZ vaccine according to different schedules is compared with the response in children who received the first dose of rMenB+OMV NZ vaccine at 4 years of age.
Time Frame: Day 31 (1 month post vaccination)
Population: Analysis was done on FAS, Immunogenicity.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48 | B48 50
Number analyzed (Participants) | 26 | 18 | 16 | 16 | 26 | 15 | 40 | 25 | 26 | 175
Percentages of subjects
  H44/76 strain; N=26,18,16,16,26,15,39,25,26,175 | 92 [75 to 99] | 100 [81 to 100] | 100 [79 to 100] | 100 [79 to 100] | 96 [80 to 100] | 93 [68 to 100] | 97 [87 to 100] | 96 [80 to 100] | 96 [80 to 100] | 63 [55 to 70]
  5/99 strain; N=26,18,16,15,25,15,38,25,26,168 | 96 [80 to 100] | 94 [73 to 100] | 94 [70 to 100] | 100 [78 to 100] | 92 [74 to 99] | 100 [78 to 100] | 97 [86 to 100] | 96 [80 to 100] | 85 [65 to 96] | 86 [80 to 91]
  NZ 98/254 strain; N=26,18,16,16,26,15,40,25,26,173 | 81 [61 to 93] | 61 [36 to 83] | 81 [54 to 96] | 69 [41 to 89] | 88 [70 to 98] | 73 [45 to 92] | 88 [73 to 96] | 72 [51 to 88] | 85 [65 to 96] | 17 [12 to 24]
  M10713 strain; N=24,17,16,12,23,15,35,24,25,158 | 38 [19 to 59] | 47 [23 to 72] | 31 [11 to 59] | 33 [10 to 65] | 39 [20 to 61] | 40 [16 to 68] | 49 [31 to 66] | 46 [26 to 67] | 32 [15 to 54] | 21 [15 to 28]

11. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥1:5 and ≥1:8 Following a Third Dose of rMenB+OMV NZ Vaccine (at 4 Years of Age), Who Had Previously Received 2 Catch up Doses of the Same Vaccine According to Different Schedules
Description: The percentages of subjects with hSBA titers ≥1:5 and hSBA titers ≥1:8 at one month after a third dose of rMenB+OMV NZ vaccine was given to children, who had previously received 2 catch up doses (at 12,14 or 18,20 or 24,26 months) of the same vaccine according to different schedules, are reported.
Time Frame: Day 31 (1 month post vaccination)
Population: Analysis was done on FAS (Immunogenicity).
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B12 14_48 | B18 20_48 | B24 26_48 | B48_50
Number analyzed (Participants) | 97 | 10 | 12 | 175
Percentages of subjects
  hSBA≥ 1:5 (H44/76 strain) | 100 [96 to 100] | 100 [69 to 100] | 100 [74 to 100] | 71 [64 to 78]
  hSBA≥ 1:5 (5/99 strain; N=95,10,12,171) | 100 [96 to 100] | 100 [69 to 100] | 100 [74 to 100] | 90 [85 to 94]
  hSBA≥ 1:5 (NZ 98/254 strain; N=95,10,12,173) | 96 [90 to 99] | 70 [35 to 93] | 100 [74 to 100] | 24 [18 to 31]
  hSBA≥ 1:5 (M10713 strain; N=90,9,10,167) | 93 [86 to 98] | 100 [66 to 100] | 90 [55 to 100] | 77 [70 to 83]
  hSBA≥ 1:8 (H44/76 strain) | 100 [96 to 100] | 100 [69 to 100] | 100 [74 to 100] | 63 [55 to 70]
  hSBA≥ 1:8 (5/99 strain; N=94,10,12,171) | 100 [96 to 100] | 100 [69 to 100] | 100 [74 to 100] | 87 [81 to 92]
  hSBA≥ 1:8 (NZ 98/254 strain; N=95,10,12,173) | 95 [88 to 98] | 60 [26 to 88] | 100 [74 to 100] | 17 [12 to 24]
  hSBA≥ 1:8 (M10713 strain; N=90,9,10,167) | 92 [85 to 97] | 100 [66 to 100] | 90 [55 to 100] | 74 [67 to 81]

12. Secondary Outcome: GMTs Following a Third Dose of rMenB+OMV NZ Vaccine in Children (at 4 Years of Age) Who Had Previously Received 2 Catch up Doses of the Same Vaccine According to Different Schedules
Description: The GMTs, one month following a third dose of rMenB+OMV NZ vaccine in 4 year old children who had previously received 2 catch up doses (at 12,14 or 18,20 or 24,26 months) of the same vaccine according to different schedules, are reported.
Time Frame: Day 31 (1 month post vaccination)
Population: Analysis was done on FAS (Immunogenicity).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B12 14_48 | B18 20_48 | B24 26_48 | B48 50
Number analyzed (Participants) | 97 | 10 | 12 | 183
Titers
  H44/76 strain | 154 [124 to 191] | 145 [76 to 277] | 211 [116 to 383] | 11 [8.51 to 14]
  5/99 strain; N= 94,10,12,171 | 1575 [1219 to 2034] | 2381 [1112 to 5095] | 3604 [1785 to 7278] | 34 [27 to 42]
  NZ 98/254 strain; N=95,10,12,173 | 31 [25 to 39] | 18 [8.87 to 35] | 47 [25 to 88] | 2.25 [1.84 to 2.75]
  M10713 strain; N=90,9,10,167 | 38 [29 to 49] | 74 [34 to 164] | 84 [39 to 180] | 20 [15 to 25]

13. Secondary Outcome: GMRs of GMTs in Children Following a Third Dose of rMenB+OMV NZ Vaccine (at 4 Years of Age) Who Previously Received 2 Catch up Doses of the Same Vaccine According to Different Schedules.
Description: The GMRs of GMTs following a third dose of rMenB+OMV NZ vaccine (one month post 3rd dose/persistence at 48 months) in children, who had previously received 2 catch up doses (at 12, 14 or 18, 20 or 24, 26 months) of the same vaccine according to different schedules, are reported.
Time Frame: Day 31 (1 month post vaccination)
Population: Analysis was done on FAS (Immunogenicity).
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | B12 14_48 | B18 20_48 | B24 26_48 | B48 50
Number analyzed (Participants) | 97 | 10 | 11 | 175
Ratio
  H44/76 strain | 99 [79 to 125] | 67 [34 to 135] | 133 [68 to 258] | 10 [8.2 to 13]
  5/99 strain; N=92,10,11,168 | 70 [57 to 86] | 51 [27 to 95] | 55 [30 to 99] | 29 [23 to 37]
  NZ 98/254 strain; N=93,10,11,173 | 27 [21 to 36] | 5.96 [2.7 to 13] | 38 [18 to 81] | 2.25 [1.84 to 2.75]
  M10713 strain; N=88,9,9,158 | 5.24 [3.91 to 7.02] | 7.06 [2.92 to 17] | 7.35 [3.03 to 18] | 2 [1.62 to 2.46]

14. Secondary Outcome: Percentages of Subjects With a 4-fold Increase in hSBA Titers Following a Third Dose of rMenB+OMV NZ Vaccine Given at 4 Years of Age to Children Who Previously Received 2 Catch up Doses of the Same Vaccine
Description: The percentage of subjects with a four-fold increase in hSBA titers following a third dose of rMenB+OMV NZ vaccine, who had previously received 2 catch up doses (at 12, 14 or 18, 20 or 24, 26 months) of rMenB+OMV NZ vaccine according to different schedules,are reported.
  Fourfold increase is defined as- for subjects with a pre-vaccination titer <1:2 to a post-vaccination titer ≥1:8 and for subjects with a pre-vaccination titer ≥1:2 to a post-vaccination titer ≥ 4 fold pre-vaccination titer.
Time Frame: Day 31 (1 month post vaccination)
Population: Analysis was done on FAS (Immunogenicity).
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B12 14_48 | B18 20_48 | B24 26_48 | B48 50
Number analyzed (Participants) | 95 | 10 | 11 | 175
Percentages of subjects
  H44/76 strain | 99 [94 to 100] | 90 [55 to 100] | 100 [72 to 100] | 63 [55 to 70]
  5/99 strain; N=92,10,11,168 | 100 [96 to 100] | 90 [55 to 100] | 100 [72 to 100] | 86 [80 to 91]
  NZ 98/254 strain; N=93,10,11,173 | 94 [86 to 98] | 50 [19 to 81] | 100 [72 to 100] | 17 [12 to 24]
  M10713 strain; N=88,9,9,158 | 58 [47 to 68] | 67 [30 to 93] | 56 [21 to 86] | 21 [15 to 28]

15. Secondary Outcome: Percentages of Subjects With hSBA ≥1:5 and ≥1:8 in Response of Two Catch up Doses of rMenB+OMV NZ Vaccine When Administered to Children at 4 Years of Age.
Description: The sufficiency of immune response is reported in terms of percentages of subjects with hSBA ≥1:5 and ≥1:8 in response of two catch up doses of rMenB+OMV NZ vaccine, administered two months apart, in children at 4 years of age.
  Immune response was considered sufficient if the lower limit of the two-sided 95% CI for the percentage of subjects achieving hSBA ≥ 1:5 at one month after the two-dose series was ≥ 70% for all three indicator (H44/76; 5/99 and NZ 98/254) strains.
  Immune sufficiency was not applicable for M10713 strain.
Time Frame: Day 91 (1 month post second vaccination)
Population: Analysis was done on FAS (Immunogenicity).
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B48_50
Number analyzed (Participants) | 175
Percentages of subjects
  hSBA≥ 1:5 (H44/76 strain) | 100 [98 to 100]
  hSBA≥ 1:5 (5/99 strain) | 100 [98 to 100]
  hSBA≥ 1:5 (NZ 98/254 strain; N=174) | 91 [85 to 95]
  hSBA≥ 1:8 (H44/76 strain) | 100 [98 to 100]
  hSBA≥ 1:8 (5/99 strain) | 100 [98 to 100]
  hSBA≥ 1:8 (NZ 98/254 strain; N=174) | 80 [73 to 86]

16. Secondary Outcome: GMTs Following 2 Catch up Doses of rMenB+OMV NZ Vaccine at 4 Years of Age
Description: The GMTs in children who received two catch up doses of rMenB+OMV NZ vaccine at 48 and 50 months of age are reported.
Time Frame: Day 91 (1 month post second vaccination)
Population: Analysis was done on FAS (Immunogenicity).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B48 50
Number analyzed (Participants) | 175
Titers
  H44/76 strain | 109 [98 to 120]
  5/99 strain | 343 [302 to 389]
  NZ 98/254 strain; N=174 | 17 [14 to 19]
  M10713 strain; N=171 | 47 [40 to 56]

17. Secondary Outcome: GMRs of GMTs Following 2 Catch up Doses of rMenB+OMV NZ Vaccine at 4 Years of Age
Description: The GMR of GMTs(one month post dose 2/baseline) in children following a two catch up dose of rMenB+OMV NZ at 48 and 50 months of age are reported.
Time Frame: Day 91 (1 month post second vaccination)
Population: Analysis was done on FAS (Immunogenicity).
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | B48 50
Number analyzed (Participants) | 175
Ratio
  H44/76 strain | 105 [94 to 116]
  5/99 strain; N=172 | 299 [256 to 350]
  NZ 98/254 strain; N=174 | 17 [14 to 19]
  M10713 strain; N=171 | 5.12 [3.95 to 6.65]

18. Secondary Outcome: Percentages of Subjects With 4-fold Increase in Serum Bactericidal Titers, Following 2 Catch up Doses of rMenB+OMV NZ Vaccine at 4 Years of Age
Description: The percentages of subjects with 4-fold increase in hSBA titers, one month following a two catch up dose of rMenB+OMV NZ at 4 years of age are reported.
Time Frame: Day 91 (1 month post second vaccination)
Population: Analysis was done on FAS (Immunogenicity).
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | B48 50
Number analyzed (Participants) | 175
Percentages of subjects
  H44/76 strain | 100 [98 to 100]
  5/99 strain; N=172 | 99 [97 to 100]
  NZ 98/254 strain; N=174 | 80 [73 to 86]
  M10713 strain; N=161 | 51 [43 to 59]

19. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After Receiving a 5th Dose of rMenB+OMV NZ Vaccine (at 4 Years of Age)
Description: The safety and tolerability of the 5th dose rMenB+OMV NZ vaccine in children (at 4 years of age) who had previously received 3 primary doses (at 2, 3, 4, or 2, 4, 6 months) followed by a booster dose (at 12, 18 or 24 months) of rMenB+OMV NZ vaccine according to different schedules in the earlier studies is reported as number of subjects with solicited local and systemic adverse events.
Time Frame: From day 1 to day 7 after vaccination
Population: Analysis was done on the safety population, ie, all subjects in the Exposed population who provided post vaccination and post-baseline safety data.
Measure: Number; unit: Number of subjects
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48
Number analyzed (Participants) | 29 | 20 | 17 | 19 | 27 | 17 | 43 | 29 | 27
Number of subjects
  Any local | 27 | 18 | 17 | 16 | 24 | 17 | 38 | 28 | 27
  Injection site Pain (mild) | 4 | 5 | 1 | 6 | 5 | 2 | 4 | 6 | 7
  Injection site Pain (moderate) | 18 | 9 | 13 | 4 | 14 | 9 | 24 | 14 | 17
  Injection site Pain (severe) | 5 | 4 | 3 | 6 | 4 | 5 | 10 | 8 | 3
  Injection site Erythema (25 - 50 mm) | 2 | 3 | 3 | 5 | 6 | 3 | 5 | 6 | 5
  Injection site Erythema (51 - 100 mm) | 5 | 2 | 1 | 2 | 7 | 3 | 10 | 6 | 3
  Injection site Erythema (>100 mm) | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
  Injection site Induration (25 - 50 mm) | 2 | 2 | 1 | 2 | 5 | 2 | 6 | 7 | 6
  Injection site Induration (51 - 100 mm) | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 1
  Injection site Induration (>100 mm) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Injection site Swelling (25 - 50 mm) | 1 | 3 | 3 | 4 | 5 | 3 | 7 | 7 | 4
  Injection site Swelling (51 - 100 mm) | 1 | 0 | 1 | 2 | 3 | 2 | 7 | 5 | 1
  Injection site Swelling (>100 mm) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Any Systemic | 26 | 15 | 14 | 18 | 19 | 13 | 36 | 27 | 23
  Change in eating habits | 12 | 6 | 6 | 12 | 7 | 8 | 20 | 11 | 13
  Rash | 2 | 1 | 0 | 5 | 2 | 4 | 7 | 5 | 2
  Arthralagia | 12 | 4 | 6 | 9 | 8 | 5 | 11 | 8 | 12
  Headache | 5 | 1 | 6 | 3 | 2 | 3 | 7 | 5 | 8
  Irritability | 18 | 9 | 11 | 14 | 13 | 8 | 23 | 20 | 16
  Diarrhea | 4 | 1 | 1 | 2 | 4 | 2 | 6 | 4 | 3
  Vomiting | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 3 | 2
  Fever (≥ 38.0 °C) | 6 | 3 | 3 | 2 | 1 | 1 | 5 | 4 | 2
  Antipyretic used (prophylactically) | 1 | 2 | 1 | 1 | 2 | 1 | 7 | 1 | 1
  Antipyretic used (therapeutically) | 5 | 5 | 4 | 3 | 3 | 1 | 10 | 4 | 3

20. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After Receiving a 3rd Dose of rMenB+OMV NZ Vaccine (at 4 Years of Age)
Description: The safety and tolerability of the 3rd dose rMenB+OMV NZ vaccine in children (at 4 years of age) who had previously received 2 catch up doses (at 12, 14 or 18, 20 or 24, 26 months) of rMenB+OMV NZ vaccine according to different schedules is reported as number of subjects with solicited local and systemic adverse events.
Time Frame: From day 1 to day 7 after vaccination
Population: Analysis was done on the safety population.
Measure: Number; unit: Number of subjects
Arm/Group | B12 14_48 | B18 20_48 | B24 26_48
Number analyzed (Participants) | 99 | 10 | 12
Number of subjects
  Any local | 94 | 9 | 11
  Injection site Pain (mild) | 33 | 2 | 2
  Injection site Pain (moderate) | 42 | 6 | 8
  Injection site Pain (severe) | 19 | 1 | 1
  Injection site Erythema (25 - 50 mm) | 12 | 2 | 0
  Injection site Erythema (51 - 100 mm) | 7 | 1 | 0
  Injection site Erythema (>100 mm) | 2 | 0 | 0
  Injection site Induration (25 - 50 mm) | 8 | 1 | 0
  Injection site Induration (51 - 100 mm) | 0 | 0 | 0
  Injection site Induration (>100 mm) | 1 | 0 | 0
  Injection site Swelling (25 - 50 mm) | 18 | 2 | 3
  Injection site Swelling (51 - 100 mm) | 2 | 0 | 1
  Injection site Swelling (>100 mm) | 0 | 0 | 0
  Any Systemic | 78 | 6 | 9
  Change in eating habits | 42 | 0 | 3
  Rash | 13 | 0 | 0
  Arthralagia | 28 | 1 | 6
  Headache | 20 | 2 | 4
  Irritability | 53 | 4 | 5
  Diarrhea | 5 | 0 | 2
  Vomiting | 6 | 2 | 1
  Fever (≥ 38.0 °C) | 16 | 4 | 5
  Antipyretic used (prophylactically) | 5 | 2 | 2
  Antipyretic used (therapeutically) | 18 | 4 | 5

21. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After Receiving a 2 Catch up Doses of rMenB+OMV NZ Vaccine at 4 Years of Age
Description: The safety and tolerability of rMenB+OMV NZ vaccine in 4 year old children who received 2 catch up doses of rMenB+OMV NZ vaccine at 48 and 50 months, is reported as number of subjects with solicited local* and systemic adverse events.
Time Frame: From day 1 to day 7 after any vaccination
Population: Analysis was done on the safety population.
Measure: Number; unit: Number of subjects
Groups:
- B48 50 (After 1st Dose); B48 50 (After 2nd Dose): Newly recruited 4 year old naive subjects who received 2 catch-up doses of rMenB+OMV NZ vaccine, two months apart, in the present study.
Arm/Group | B48 50 (After 1st Dose) | B48 50 (After 2nd Dose)
Number analyzed (Participants) | 205 | 194
Number of subjects
  Any local | 186 | 161
  Injection site Pain (mild) | 81 | 70
  Injection site Pain (moderate) | 77 | 66
  Injection site Pain (severe) | 27 | 21
  Injection site Erythema (25 - 50 mm; N= 204, 194) | 34 | 15
  Injection site Erythema (51 - 100 mm; N= 204, 194) | 8 | 19
  Injection site Erythema (>100 mm; N= 204, 194) | 1 | 0
  Injection site Induration (25 - 50 mm; N= 204, 194 | 23 | 16
  Injection site Induration (51-100 mm; N= 204, 194) | 3 | 4
  Injection site Induration(>100 mm; N= 204, 194 | 0 | 0
  Injection site Swelling (25 - 50 mm; N= 204, 194 | 26 | 20
  Injection site Swelling (51 - 100 mm; N= 204, 194) | 3 | 4
  Injection site Swelling (>100 mm; N= 204, 194) | 1 | 0
  Any Systemic | 137 | 108
  Rash; N=201, 192 | 15 | 10
  Change in eating habits; N= 203, 194 | 49 | 43
  Headache; N= 204, 194 | 25 | 24
  Arthralagia; N= 203, 192 | 45 | 40
  Irritability; N= 204, 193 | 67 | 58
  Vomiting | 8 | 6
  Diarrhea; N= 204, 193 | 11 | 8
  Fever (≥ 38.0 °C; N= 204, 189) | 20 | 16
  Antipyretic used (prophylactically; N= 204, 193) | 17 | 23
  Antipyretic used (therapeutically; N= 204, 193) | 22 | 24

22. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs After Receiving a 5th Dose of rMenB+OMV NZ Vaccine (at 4 Years of Age)
Description: The safety and tolerability of the 5th dose rMenB+OMV NZ vaccine in children (at 4 years of age) who had previously received 3 primary doses (at 2, 3, 4,or 2, 4, 6 months) followed by a booster dose (at 12, 18 or 24 months) of rMenB+OMV NZ vaccine according to different schedules in the earlier studies is reported as number of subjects with unsolicited AEs, Serious Adverse Events (SAE), AEs leading to premature withdrawal.
Time Frame: From day 1 to study termination
Population: Analysis was done on the safety population.
Measure: Number; unit: Number of subjects
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48
Number analyzed (Participants) | 30 | 20 | 17 | 19 | 27 | 17 | 43 | 29 | 28
Number of subjects
  Any AEs | 8 | 4 | 4 | 7 | 7 | 3 | 11 | 11 | 6
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs leading to withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs After Receiving a 3rd Dose of rMenB+OMV NZ Vaccine (at 4 Years of Age)
Description: The safety and tolerability of the 3rd dose rMenB+OMV NZ vaccine in children (at 4 years of age) who had previously received 2 catch up doses (at 12, 14 or 18, 20 or 24, 26 months) of rMenB+OMV NZ vaccine according to different schedules is reported as number of subjects with Unsolicited AEs, Serious Adverse Events (SAEs), AEs leading to premature withdrawal.
Time Frame: From day 1 to study termination
Population: Analysis was done on the safety population.
Measure: Number; unit: Number of subjects
Arm/Group | B12 14_48 | B18 20_48 | B24 26_48
Number analyzed (Participants) | 100 | 11 | 12
Number of subjects
  Any AE | 25 | 2 | 4
  SAEs | 0 | 0 | 0
  AEs leading to withdrawal | 0 | 0 | 0

24. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs After Any Vaccination.
Description: as for outcome 23
Time Frame: From day 1 to study termination
Population: Analysis was done on the safety population.
Measure: Number; unit: Number of participants
Arm/Group | B48 50
Number analyzed (Participants) | 206
Number of participants
  Any AEs | 105
  SAEs | 3
  AEs leading to premature withdrawal | 1

ADVERSE EVENTS:
Time Frame: Solicited local and systemic AEs, medically attended fever, use of antipyretics and all AEs were recorded for 7 days after vaccination. Serious AEs, medically attended AEs, AEs leading to withdrawal were recorded throughout the study period.
Description: Solicited AEs were collected through systematic assessment, unsolicited AEs were collected through non-systematic assessment. Number of participants at risk in groups, B+R246_12_48, B+R246_18_48, B+R246_24_48, B246_12_48, B246_18_48, B246_24_48 si referred to the subsect of subjects who actually received vaccination in the present study.
Arm/Group | B+R246_12_48 | B+R246_18_48 | B+R246_24_48 | B246_12_48 | B246_18_48 | B246_24_48 | B+R234_12_48 | B+R234_18_48 | B+R234_24_48 | B12 14_48 | B18 20_48 | B24 26_48 | B48 50
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/20 | 0/17 | 0/19 | 0/27 | 0/17 | 0/43 | 0/29 | 0/28 | 0/100 | 0/11 | 0/12 | 3/206
Other Adverse Events (participants affected / at risk) | 29/30 | 19/20 | 17/17 | 18/19 | 25/27 | 17/17 | 42/43 | 28/29 | 27/28 | 97/100 | 10/11 | 12/12 | 200/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B+R246_12_48 (N=30) | B+R246_18_48 (N=20) | B+R246_24_48 (N=17) | B246_12_48 (N=19) | B246_18_48 (N=27) | B246_24_48 (N=17) | B+R234_12_48 (N=43) | B+R234_18_48 (N=29) | B+R234_24_48 (N=28) | B12 14_48 (N=100) | B18 20_48 (N=11) | B24 26_48 (N=12) | B48 50 (N=206)
CROUP INFECTIOUS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B+R246_12_48 (N=30) | B+R246_18_48 (N=20) | B+R246_24_48 (N=17) | B246_12_48 (N=19) | B246_18_48 (N=27) | B246_24_48 (N=17) | B+R234_12_48 (N=43) | B+R234_18_48 (N=29) | B+R234_24_48 (N=28) | B12 14_48 (N=100) | B18 20_48 (N=11) | B24 26_48 (N=12) | B48 50 (N=206)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
INJECTION SITE ERYTHEMA (General disorders) | 23 | 13 | 13 | 16 | 21 | 14 | 38 | 24 | 23 | 73 | 8 | 7 | 166
INJECTION SITE INDURATION (General disorders) | 21 | 8 | 11 | 14 | 11 | 12 | 24 | 21 | 19 | 46 | 6 | 4 | 117
INJECTION SITE PAIN (General disorders) | 27 | 19 | 17 | 16 | 23 | 16 | 38 | 28 | 27 | 94 | 9 | 11 | 192
INJECTION SITE SWELLING (General disorders) | 12 | 7 | 10 | 13 | 10 | 11 | 25 | 17 | 14 | 46 | 6 | 7 | 96
PYREXIA (General disorders) | 7 | 3 | 3 | 2 | 1 | 1 | 7 | 4 | 2 | 19 | 5 | 5 | 36
ACUTE TONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
EAR INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 6
ERYTHEMA INFECTIOSUM (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3
SOMNOLENCE (Nervous system disorders) | 18 | 7 | 8 | 9 | 12 | 6 | 22 | 21 | 14 | 52 | 3 | 3 | 105
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 11
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 5 | 2 | 4 | 7 | 5 | 2 | 13 | 0 | 0 | 24
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 | 4 | 6 | 9 | 8 | 5 | 11 | 8 | 12 | 28 | 1 | 6 | 67
HEADACHE (Nervous system disorders) | 5 | 1 | 6 | 3 | 2 | 3 | 7 | 5 | 8 | 20 | 2 | 4 | 40
EATING DISORDER (Psychiatric disorders) | 12 | 6 | 6 | 12 | 7 | 8 | 20 | 11 | 13 | 42 | 0 | 3 | 75
IRRITABILITY (Psychiatric disorders) | 18 | 9 | 11 | 14 | 13 | 8 | 23 | 20 | 16 | 53 | 4 | 5 | 91
CATARRH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.